CLINICAL TRIAL: NCT03937245
Title: Epidemiology and Determinants of Outcomes of Hospital Acquired Blood Stream Infections in the Intensive Care: the Eurobact II Multinational Cohort Study
Brief Title: Epidemiology and Determinants of Outcomes of Hospital Acquired Blood Stream Infections in the Intensive Care
Acronym: EurobactII
Status: Completed | Type: Observational
Sponsor: Outcome Rea (Other)
Collaborators: European Society of Intensive Care Medicine (Other); European Society of Clinical Microbiology and Infectious Diseases (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: EurobactII
Record Dates: First submitted 2019-05-01; First posted 2019-05-03 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Bacteremia; Sepsis; Hospital Acquired Condition; Resistance Bacterial
Keywords: Hospital-acquired infection; Blood stream infection; Bacteremia; Intensive care
MeSH Terms: conditions — Bacteremia; Sepsis; Iatrogenic Disease; Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HA-BSI: Patients with HA-BSI treated in an ICU

SUMMARY:
Eurobact II will investigate the mortality and morbidity of hospital-acquired blood stream infections in patients treated in intensive care units (ICU). It will investigate the effects of the micro-organism and its characteristics, such as type and resistance to antibiotics on the infection and its consequences. It will also investigate the effects of the antibiotics and other treatments on survival of patients. Eurobact II will include patients from multiple ICUs in multiple countries.

DETAILED DESCRIPTION:
Eurobact II is a multinational multicentre cohort study that will include patients with hospital-acquired blood stream infections (HA-BSI) treated in ICUs around the globe. It will provide with an update of the epidemiology of HA-BSI since the Eurobact I study. It is designed to investigate the effects of HA-BSI on mortality at day 28. To describe the determinants of outcomes of HA-BSI, specifically the effects of the source of infection, the microorganism, the characteristics of antimicrobial therapy and of source control. It will investigate patient specific and organizational factors and will describe the determinants of management of HA-BSI in ICUs.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 Years.
* Hospital Acquired Bloodstream Infection (HA-BSI).
* Treated in the ICU.

  * ICU acquired OR
  * Hospital acquired prior to ICU admission

Exclusion Criteria:

* Patients that had a positive blood culture in the hospital and transferred to ICU for a different reason than specific treatment of the causes or consequences of HA-BSI.
* Previous inclusion in the study.

  * HA-BSI is defined as a positive blood culture (BC) sampled after 48 hours following hospital admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a HA-BSI treated in an ICU
Sampling Method: Non-Probability Sample
Enrollment: 3058 (Actual)
Dates: Start 2019-08-30 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-03 (Actual)

PRIMARY OUTCOMES:
Mortality | 28 days
  Vital status

SECONDARY OUTCOMES:
Progress of organ failures | 7 days
  Assessed by the components of the SOFA score
Days free or organ supportive therapy | 28 days
  Days free of renal replacement therapy, mechanical ventilation, vasopressors, intensive care unit
Clinical cure | 7 days, 28 days
  As evaluated by the treating clinician
Microbiological cure | 7 days, 28 days
  Presence of persisting or relapsing blood stream infection

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Tabah, MD, Principal Investigator — ICU, Redcliffe Hospital, Faculty of Medicine, UQ, Brisbane, QLD, Australia.; Jean-Francois Timsit, MD,PhD, Study Director — Medical and infectious diseases ICU, Bichat hospital, IAME U 1137,Paris,France
Locations (2):
- Redcliffe Hospital, Brisbane, Queensland, Australia
- Reanimation Medicale et Infectieuse-Hopital Bichat, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tabah A, Koulenti D, Laupland K, Misset B, Valles J, Bruzzi de Carvalho F, Paiva JA, Cakar N, Ma X, Eggimann P, Antonelli M, Bonten MJ, Csomos A, Krueger WA, Mikstacki A, Lipman J, Depuydt P, Vesin A, Garrouste-Orgeas M, Zahar JR, Blot S, Carlet J, Brun-Buisson C, Martin C, Rello J, Dimopoulos G, Timsit JF. Characteristics and determinants of outcome of hospital-acquired bloodstream infections in intensive care units: the EUROBACT International Cohort Study. Intensive Care Med. 2012 Dec;38(12):1930-45. doi: 10.1007/s00134-012-2695-9. Epub 2012 Sep 26. PMID 23011531
- [Derived] Gajdos L, Buetti N, Tabah A, Ruckly S, Akova M, Sjoval F, Arvaniti K, de Waele J, Bracht H, Barbier F, Timsit JF; EUROBACT-2 Study Group, the European Society of Intensive Care Medicine (ESICM), the European Society of Clinical Microbiology, the Infectious Diseases (ESCMID) Study Group for Infections in Critically Ill Patients (ESGCIP) and the OUTCOMEREA Network. Shortening antibiotic therapy duration for hospital-acquired bloodstream infections in critically ill patients: a causal inference model from the international EUROBACT-2 database. Intensive Care Med. 2025 Mar;51(3):518-528. doi: 10.1007/s00134-025-07857-6. Epub 2025 Apr 7. PMID 40192823
- [Derived] Buetti N, Tabah A, Loiodice A, Ruckly S, Aslan AT, Montrucchio G, Cortegiani A, Saltoglu N, Kayaaslan B, Aksoy F, Murat A, Akdogan O, Saracoglu KT, Erdogan C, Leone M, Ferrer R, Paiva JA, Hayashi Y, Ramanan M, Conway Morris A, Barbier F, Timsit JF; Eurobact 2 study group. Different epidemiology of bloodstream infections in COVID-19 compared to non-COVID-19 critically ill patients: a descriptive analysis of the Eurobact II study. Crit Care. 2022 Oct 18;26(1):319. doi: 10.1186/s13054-022-04166-y. PMID 36258239
- See also: Eurobact II website — http://www.eurobact.org

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-19): https://cdn.clinicaltrials.gov/large-docs/45/NCT03937245/Prot_SAP_000.pdf